CLINICAL TRIAL: NCT01892748
Title: Effects of Cholecalciferol Supplementation on Disease Activity, Fatigue and Bone Mass on Juvenile Onset Systemic Lupus Erythematosus.
Brief Title: Cholecalciferol Supplementation on Disease Activity, Fatigue and Bone Mass on Juvenile Systemic Lupus Erythematosus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ROSA MARIA RODRIGUES PEREIRA (Other)
Responsible Party: Sponsor-Investigator, ROSA MARIA RODRIGUES PEREIRA, Associate Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VITD59/11
Record Dates: First submitted 2013-06-17; First posted 2013-07-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Juvenile; Cholecalciferol; Disease activity; Bone Mass; Fatigue; Safety
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol 50.000IU/week (Active Comparator): patients will receive vitamin D3 (50.000 IU/week) for 24weeks
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): patients receive placebo in similar capsules of cholecalciferol for 24weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — All patients and physicians were blinded to group assignment and treatment allocation. The first group received oral cholecalciferol of 50,000 IU/week and for 6 months. All subjects were evaluated at baseline and after the end of supplementation for clinical and laboratory parameters.
  Other Names: Vitamin D3
  Arms: Cholecalciferol 50.000IU/week
Drug: Placebo — The second group received identical placebo tablets for 6 months. All subjects were evaluated at baseline and after the end of supplementation for clinical and laboratory parameters.
  Other Names: No other names
  Arms: Placebo

SUMMARY:
The potential role of vitamin D on disease susceptibility, activity and severity has been considered for several autoimmune rheumatologic diseases include systemic lupus erythematosus (SLE) . Although, there are few studies of vitamin D supplementation in SLE patients, especially in Juvenile Onset Systemic Lupus Erythematosus (JoSLE).

The objective of this study is to evaluate the effect of vitamin D supplementation (cholecalciferol 50.000 international units (IU)/week for 24 weeks) on disease activity (clinical and laboratory parameters), fatigue and bone mass.

DETAILED DESCRIPTION:
This is a study 24-week, two arm, double blinded randomized clinical trial to evaluate the effects of high-dose vitamin D3 supplementation compared with placebo, on activity disease, fatigue and bone mass.

Sixty JoSLE patients will be randomized to receive placebo or vitamin D3 (50.000 IU/week) for 24weeks. The patients return to visits in week 12 and week 24 for evaluation. Study will record clinical history, drugs in use, disease activity, and bone mass parameters.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed
* 4 of the 11 modified American College of Rheumatology (ACR) Revised Criteria for the Classification of Systemic Lupus Erythematosus .
* SLEDAI < 8 at Screening and at Baseline
* Stable immunosuppressive dose prior to randomization.
* Body Mass Index < 30
* Able to swallow pills at randomization

Exclusion Criteria:

* Refuse of the patient or the legal responsible
* Use of vitamin D2 or D3 supplementation
* Significant renal insufficiency
* Primary hyperparathyroidism (known)
* History of nephrolithiasis (known)
* Diabetes mellitus requiring insulin therapy
* History of vertebral compression fractures (known)
* Pregnancy
* Use of bisphosphonates

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The change in Disease Activity Score (SLEDAI) | baseline to week 12 and 24

SECONDARY OUTCOMES:
The change in Fatigue Score | baseline to week 12 and 24
The change in Bone Mineral Parameters | baseline to week 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Rosa MR Pereira, MD PhD, Principal Investigator — University of Sao Paulo - School of Medicine; Glauce L Lima, MD, Study Chair — University of Sao Paulo - School of Medicine
Locations (1):
- University of Sao Paulo - School of Medicine, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lima GL, Paupitz JA, Aikawa NE, Alvarenga JC, Pereira RMR. A randomized double-blind placebo-controlled trial of vitamin D supplementation in juvenile-onset systemic lupus erythematosus: positive effect on trabecular microarchitecture using HR-pQCT. Osteoporos Int. 2018 Mar;29(3):587-594. doi: 10.1007/s00198-017-4316-5. Epub 2017 Nov 19. PMID 29152675
- [Derived] Lima GL, Paupitz J, Aikawa NE, Takayama L, Bonfa E, Pereira RM. Vitamin D Supplementation in Adolescents and Young Adults With Juvenile Systemic Lupus Erythematosus for Improvement in Disease Activity and Fatigue Scores: A Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Care Res (Hoboken). 2016 Jan;68(1):91-8. doi: 10.1002/acr.22621. PMID 25988278